CLINICAL TRIAL: NCT01630928
Title: Renal Sympathetic Denervation for Treatment Resistant Hypertension and Potential Effects on Glucose Metabolism and Cardiovascular Risk-Factors (The Re-Shape CV-Risk Study)
Brief Title: Renal Sympathetic Denervation and Potential Effects on Glucose Metabolism and Cardiovascular Risk-Factors
Acronym: Re-Shape
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: University of Tromso (Other); The Royal Norwegian Ministry of Health (Other); Odd Berg Medical research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/1296 (REK)
Record Dates: First submitted 2012-06-26; First posted 2012-06-28 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Hypertension, Resistant to Conventional Therapy
Keywords: Renal denervation; Resistant Hypertension; Cardiovascular disease; Diabetes; Quality of LIfe
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Renal sympathetic denervation (Experimental): Patients with treatment resistant hypertension
  Interventions: Procedure: Renal sympathetic denervation

INTERVENTIONS:
Procedure: Renal sympathetic denervation — This is a mini-invasive trans-catheter procedure with access via a 6F introducer in one of the femoral arteries. The renal sympathetic nerves arise from T10-L2, arborize around the renal artery and primarily lie within the adventitia. A specialized radiofrequency (RF) ablation catheter is introduced into the renal arteries, first one side, then on the other. Usually, 4-6 two-minute treatments per artery using a proprietary RF generator with automated low power and built-in safety algorithms are sufficient to ablate the sympathetic afferent and efferent fibers.
  Other Names: Symplicity Catheter (Medtronic)

SUMMARY:
The Re-Shape CV-Risk Study is a clinical study where renal adrenergic denervation (RDN) is done in high risk patients with treatment-resistant hypertension. RDN is a mini-invasive, percutaneous technique where an ablation catheter is inserted through a femoral artery into the renal arteries, for destruction of the adrenergic nerve bundles in the artery adventitia by means of radio-frequency ablation. RDN leads to sympathetic denervation of the kidneys, which in the "Symplicity trials" led to an impressive reduction of blood pressure (- 33 /-11 mmHg). In a pilot study, where 40 % of the patients had diabetes, RDN seemed to have beneficial effects not only on blood pressure, but also on insulin sensitivity and hyperinsulinaemia.

The investigators aim to introduce RDN as a clinical study where blood pressure reduction and methodical, technical aspects will be evaluated, but more importantly, also additional effects of RDN on sub-clinical organ damage (endothelial function, vascular stiffness, fundus-, heart-, kidney injury), quality of life, arrhythmia, and glucose metabolism. The investigators hypothesis is that RDN will have positive effect on glucose metabolism, QOL and sub-clinical organ damage.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 Years.
* Resistant hypertension, as defined in the 2007 ESH-ESC guidelines and confirmed by ambulatory or home blood pressure measurements. (Here office BP > 140/90 mmHg on 4 or more antihypertensive drugs in adequate dosages (including one diuretic) or certified drug intolerance).
* No known secondary reason for hypertension
* Negative pregnancy test (preferably blood hCG) for female patients of childbearing potential
* Estimated GFR (glomerular filtration rate) > 45 mL/min/1.73m².
* Willing and able to comply with follow-up requirements
* Signed informed consent

Exclusion Criteria:

* Type 1 and type 2 diabetes
* Pregnancy
* Allergy to the contrast medium used during RDN and Iohexol clearance.
* Age > 68 years
* Hemodynamically significant heart valve disease
* Pacemaker or ICD
* Medication that may interfere with the procedure (Anticoagulation, Platelet inhibitors, Steroids), if they cannot be temporarily reduced or stopped.
* Cancer
* Patients with transplanted kidneys
* Reno vascular conditions like diameter < 4mm, renal artery stenosis or significant atherosclerosis, previous renal artery stenting

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | from baseline to six months
  Change in blood pressure from baseline to six months after the intervention
Change in blood pressure | from baseline to two years
  Change in blood pressure from baseline to two years after the intervention

SECONDARY OUTCOMES:
Change in quality of Life | From baseline to six months
  The international questionnaires SF-36 and 15-D, with some additional specific questions previously used in international studies will be used for evaluation of RDN effect on symptoms and QOL.
Changes in glucose production and insulin sensitivity | from baseline to six months
  Glucose metabolism will be assessed with oral glucose tolerance test and 2-step euglycemic, hyperinsulinaemic clamp with tracer technique (6,6-2H2-glucose + HOTGINF / measurement of tracer-to-tracee ratio with mass spectrometry): Assessment of endogenous glucose production at fasting condition, at insulin levels around 30 mU/ml (hepatic insulin sensitivity), and at insulin levels of 65-68 mU/ml, imitating the postprandial state (peripheral insulin resistance). Assessment of glucose uptake at these conditions (insulin sensitivity).
Change in quality of Life | From baseline to two years
  The international questionnaires SF-36 and 15-D, with some additional specific questions previously used in international studies will be used for evaluation of RDN effect on symptoms and QOL.
Changes in glucose production and insulin sensitivity | from baseline to two years
  Glucose metabolism will be assessed with oral glucose tolerance test and 2-step euglycemic, hyperinsulinaemic clamp with tracer technique (6,6-2H2-glucose + HOTGINF / measurement of tracer-to-tracee ratio with mass spectrometry): Assessment of endogenous glucose production at fasting condition, at insulin levels around 30 mU/ml (hepatic insulin sensitivity), and at insulin levels of 65-68 mU/ml, imitating the postprandial state (peripheral insulin resistance). Assessment of glucose uptake at these conditions (insulin sensitivity).
Effect of RDN on subclinical organ injury: Myocardium | from baseline to six months
  Long standing hypertension leads to sub-clinical organ damage:
  Myocardial and vascular remodeling measured with echo cardiography. Wall stiffness, left ventricular function, hypertrophy and mass.
Effect of RDN on subclinical organ injury: Myocardium | from baseline to two years
  Long standing hypertension leads to sub-clinical organ damage:
  Myocardial and vascular remodeling measured with echo cardiography. Wall stiffness, left ventricular function, hypertrophy and mass.
Effect of RDN on subclinical organ injury: Retinal vessels | from baseline to six months
  Long standing hypertension leads to sub-clinical organ damage:
  Changes in the microcirculatory vasculature detectable as early changes in retinal vascular caliber or presence of hypertensive retinopathy. High resolution photography (Carl Zeiss Meditec.) and optic coherence tomography of the retina give a direct view to microcirculation. Analyzes will be performed using computer assisted morphometry (IVAN/Retinal Analysis software. Fundus Reading center, University of Wisconsin, Madison USA).
Effect of RDN on subclinical organ injury: Retinal vessels | from baseline to two years
  Long standing hypertension leads to sub-clinical organ damage:
  Changes in the microcirculatory vasculature detectable as early changes in retinal vascular caliber or presence of hypertensive retinopathy. High resolution photography (Carl Zeiss Meditec.) and optic coherence tomography of the retina give a direct view to microcirculation. Analyzes will be performed using computer assisted morphometry (IVAN/Retinal Analysis software. Fundus Reading center, University of Wisconsin, Madison USA).
Effect of RDN on subclinical organ injury: Kidneys | from baseline to six months
  Long standing hypertension leads to sub-clinical organ damage:
  Renal dysfunction. We will measure serum creatinine, cystatin C, GFR (iohexol clearance), albumine/creatinine ratio and N-Acetyl-ß-glucosaminidase (NAG) in morning urine (two different days) before and after RDN. NAG excretion is a sign of tubular injury.
Effect of RDN on subclinical organ injury: Kidneys | from baseline to two years
  Long standing hypertension leads to sub-clinical organ damage:
  Renal dysfunction. We will measure serum creatinine, cystatin C, GFR (iohexol clearance), albumine/creatinine ratio and N-Acetyl-ß-glucosaminidase (NAG) in morning urine (two different days) before and after RDN. NAG excretion is a sign of tubular injury.
Effect of RDN on subclinical organ injury: Endothelial function | from baseline to six months
  Long standing hypertension leads to sub-clinical organ damage:
  Impaired endothelial function; assessed with plethysmography under reactive hyperemia + markers of endothelial dysfunction; Peripheral vasodilator function is measured by digital pulse amplitude tonometry using EndoPAT 2000 (Itamar Medical Ltd., Caesarea, Israel). Reactive hyperemia is produced by applying a blood pressure cuff for 5 min at a pressure of 60 mmHg higher than the systolic pressure on the upper part of the arm.
Effect of RDN on subclinical organ injury: Endothelial function | from baseline to two years
  Long standing hypertension leads to sub-clinical organ damage:
  Impaired endothelial function; assessed with plethysmography under reactive hyperemia + markers of endothelial dysfunction; Peripheral vasodilator function is measured by digital pulse amplitude tonometry using EndoPAT 2000 (Itamar Medical Ltd., Caesarea, Israel). Reactive hyperemia is produced by applying a blood pressure cuff for 5 min at a pressure of 60 mmHg higher than the systolic pressure on the upper part of the arm.
Effect of RDN on subclinical organ injury: Impedance cardiography | from baseline to two years
  Increased central blood pressure measured in ascending aorta, in addition to "augmentation index" (peak aortic pressure increase/pulse pressure) as a measure of vessel compliance, are independent predictors for hypertensive organ injury (brain, heart, kidneys). Aortic wall-stiffness (compliance) and pulse wave reflection are important determinants for central blood pressure and are among the parameters we indirectly will get from impedance cardiography (Hotman System, HEMO SAPIENS INC, Bucharest, Romania)
Effect of RDN on subclinical organ injury: Impedance cardiography | from baseline to six months
  Increased central blood pressure measured in ascending aorta, in addition to "augmentation index" (peak aortic pressure increase/pulse pressure) as a measure of vessel compliance, are independent predictors for hypertensive organ injury (brain, heart, kidneys). Aortic wall-stiffness (compliance) and pulse wave reflection are important determinants for central blood pressure and are among the parameters we indirectly will get from impedance cardiography (Hotman System, HEMO SAPIENS INC, Bucharest, Romania)

CONTACTS AND LOCATIONS:
Overall Officials: Terje K. Steigen, MD, PhD, Principal Investigator — Dept. of Cardiology, University Hospital of North Norway and University of Tromsø, Norway; Ingrid Toft, MD, PhD, Study Chair — Dept. of Nephrology, University Hospital of North Norway and University of Tromsø; Marit D Solbu, MD, PhD, Study Director — Dept of Nephrology, University Hospital of North Norway and University of Tromsø
Locations (1):
- University Hospital of North Norway, Tromsø, Norway

REFERENCES:
- [Derived] Hanssen TA, Subbotina A, Miroslawska A, Solbu MD, Steigen TK. Quality of life following renal sympathetic denervation in treatment-resistant hypertensive patients: a two-year follow-up study. Scand Cardiovasc J. 2022 Dec;56(1):174-179. doi: 10.1080/14017431.2022.2084562. PMID 35686551
- [Derived] Miroslawska AK, Gjessing PF, Solbu MD, Fuskevag OM, Jenssen TG, Steigen TK. Renal Denervation for Resistant Hypertension Fails to Improve Insulin Resistance as Assessed by Hyperinsulinemic-Euglycemic Step Clamp. Diabetes. 2016 Aug;65(8):2164-8. doi: 10.2337/db16-0205. Epub 2016 May 31. PMID 27246911